CLINICAL TRIAL: NCT01906996
Title: Comparison of Subjective, Radiological and Functional Results After Proximal Row Carpectomy and Four Corner Fusion
Brief Title: Proximal Row Carpectomy Versus Four Corner Fusion
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Daniel Herren, Dr. med., Schulthess Klinik
Other Study IDs: PRC01
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Wrist Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- proximal row carpectomy: patients were treated with a proximal row carpectomy
  Interventions: Procedure: proximal row carpectomy
- four corner fusion: patients were treated with a four corner fusion
  Interventions: Procedure: four corner fusion

INTERVENTIONS:
Procedure: proximal row carpectomy — excision of the scaphoid, lunate and triquetrum
  Groups: proximal row carpectomy
Procedure: four corner fusion — excision of the scaphoid and stiffening of the lunate, capitate and triquetrum by a plate
  Groups: four corner fusion

SUMMARY:
There are two types of interventions to treat a post-traumatic wrist osteoarthritis: the proximal row carpectomy and the four corner fusion. They are used to reduce pain and to maintain the mobility. In previous studies are shown that the proximal row carpectomy shows a better mobility of the wrist postoperatively, whereas the four corner fusion has lower progression of radiocarpale osteoarthritis.

The purpose of this study is to compare the clinical, radiological and subjective outcomes after the treatment with a proximal row carpectomy or a four corner fusion.

DETAILED DESCRIPTION:
Two surgical procedures are used to treat a post-traumatic wrist osteoarthritis, especially after scaphoid non-union advanced collapse (SNAC) and scapholunate advanced collapse (SLAC): the proximal row carpectomy and the four corner fusion. Both surgical procedures are rescue operations. They are used to reduce pain and to maintain the mobility, compared to a complete stiffening of the wrist.

In previous studies are shown that the proximal row carpectomy shows a better mobility of the wrist postoperatively and a lower complication rate, whereas the four corner fusion has a lower progression of radiocarpale osteoarthritis and a better grip strength.

The purpose of this study is to compare the clinical, radiological and subjective outcomes after the treatment with a proximal row carpectomy or a four corner fusion.

ELIGIBILITY:
Inclusion Criteria:

* post-traumatic wrist osteoarthritis
* treated with a proximal row carpectomy or four corner fusion
* signed written informed consent

Exclusion Criteria:

* no knowledge of German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a post-traumatic wrist osteoarthritis, who are treated with a proximal row carpectomy or a four corner fusion
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Range of motion of the wrist | participants will be followed up by an expected average of 4.5 years
  measurements of flexion/extension,supination/pronation and radial-/ulnarduction of the wrist

SECONDARY OUTCOMES:
complication rate | participants will be followed up by an expected average of 4.5 years
  Detection of complications of both surgical procedures

OTHER OUTCOMES:
grip strength | participants will be followed up by an expected average of 4.5 years
  measurement of grip strength
Patient-Rated Wirst Evaluation (PRWE) | participants will be followed up by an expected average of 4.5 years
  Comparison of proximal row carpectomy and four corner fusion in respect to PRWE
Michigan Hand Outcomes Questionnaire (MHQ) | participants will be followed up by an expected average of 4.5 years
  Comparison of proximal row carpectomy and four corner fusion in respect to MHQ
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | participants will be followed up by an expected average of 4.5 years
  Comparison of proximal row carpectomy and four corner fusion in rsespect to QuickDASH
Detection of radiological parameters | participants will be followed up by an expected average of 4.5 years
  Detection of arthrosis fossa lunata, impingement and loosening

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Herren, Dr. med., Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland